CLINICAL TRIAL: NCT07107919
Title: Multimodal Imaging Assessment of Chronic Kidney Disease Patients at Different Stages From a Cardio-Renal Interaction Perspective
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: QYFYEC2025-103
Record Dates: First submitted 2025-07-31; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease; Cardiac Magnetic Resonance; 18F-FAPI
Keywords: CKD; Cardiac Magnetic Resonance; 18F-FAPI
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group I (CKD stages 1-3): eGFR ≥ 30 mL/min/1.73 m²
  Interventions: Other: 18F PET/MR
- Group II (CKD stages 4-5): eGFR < 30 mL/min/1.73 m²
  Interventions: Other: 18F PET/MR

INTERVENTIONS:
Other: 18F PET/MR — Tracer: ^18F FAPI 04 is used in this study. A single intravenous bolus dose of 3.70-4.44 MBq/kg is administered.
  • Simultaneous PET/MR Acquisition: During PET imaging, cardiac MR (CMR) is performed in the supine position. All images are acquired with ECG gating and respiratory gating, during end expiratory breath holds.
  1. Cardiac Morphology and Function (Localization & Cine):Assess cardiac structure and global/regional function
  2. T2 Weighted Fat Suppressed Imaging:Evaluate myocardial edema
  3. First Pass Perfusion Imaging:Quantitatively assess the extent and severity of myocardial perfusion defects
  4. Late Gadolinium Enhancement (LGE): Detect and quantify myocardial necrosis and fibrosis
  5. T1 Mapping (Pre and Post Contrast): Quantify myocardial interstitial fibrosis
  6. T2 Mapping (Pre Contrast):Quantify myocardial edema
  7. Cardiac PET Imaging:Evaluate myocardial fibrosis characteristics using ^18F FAPI PET data

SUMMARY:
This study is a prospective cohort investigation in which consecutive eligible patients undergo 18F-FAPI PET/MR imaging. Chronic kidney disease (CKD) participants are stratified into two groups:Group I ：CKD stages 1-3（eGFR ≥ 30 mL/min/1.73 m²）,Group II :CKD stages 4-5(eGFR < 30 mL/min/1.73 m²).

Using 18F-FAPI PET/MR, we will evaluate global cardiac functional impairment and myocardial fibrosis characteristics, and analyze their associations with the degree of renal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years, regardless of sex.
2. Clinically diagnosed with chronic kidney disease (CKD), based on KDIGO guidelines.
3. Complete clinical data available.
4. Written informed consent for participation and for undergoing 18F-FAPI PET/MR imaging is obtained from the patient or their legal guardian.
5. Female participants must agree to use effective contraception during the study and for at least 6 months after its completion (e.g., sterilization, intrauterine hormonal devices, condoms, hormonal contraceptives, abstinence, or vasectomized partner). Male participants must also agree to use contraception during the study and for 6 months after its completion.

Exclusion Criteria:

1. Women who are planning to conceive, currently pregnant, or breastfeeding.
2. Contraindications to PET/MR imaging, including but not limited to metal implants, claustrophobia, or inability to tolerate cardiac MRI due to respiratory difficulties.
3. History of allergy or hypersensitivity to gadolinium-based contrast agents.
4. Presence of malignant tumors or other serious progressive diseases.
5. Patients with severe cardiac conditions, such as advanced heart failure, severe valvular disease, or cardiomyopathies.
6. Hemodynamic instability.
7. Presence of severe systemic or localized infections, or other serious comorbid conditions.
8. Incomplete clinical data.
9. Any other reason deemed by the investigators to make the subject unsuitable for participation, including inability or unwillingness to comply with study procedures and requirements.
10. Determined by the investigators to be inappropriate for inclusion in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 80 years with clinically diagnosed chronic kidney disease (CKD), classified according to the KDIGO guidelines. Participants will be stratified into two groups based on renal function: Group I (CKD stages 1-3, eGFR ≥ 30 mL/min/1.73 m²) and Group II (CKD stages 4-5, eGFR < 30 mL/min/1.73 m²). Subjects will be consecutively recruited from the Department of Nephrology and Cardiology of The Affiliated Hospital of Qingdao University. Both male and female patients will be included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Myocardial fibrosis burden measured by 18F-FAPI PET/MR | At baseline (within 1 week of enrollment)
  Myocardial uptake of 18F-FAPI quantified using SUVmax and SUVmean values from PET imaging.
Myocardial fibrosis burden measured by 18F-FAPI PET/MR | At baseline (within 1 week of enrollment)
  Native T1 value, ECV, and LGE assessed by cardiac MRI to evaluate myocardial fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Pei Nie, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No